CLINICAL TRIAL: NCT05340972
Title: Evaluate the Predictive Impact of the Meessi MEESSI Score for the Risk Stratification of Patients Admitted for Acute Heart Failure in Emergency Department
Brief Title: Evaluate the Predictive Impact of the MEESSI Score
Acronym: MEESSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Pr.Semir Nouira chef of emergency deparment, University of Monastir
Other Study IDs: MEESSI 2022
Record Dates: First submitted 2022-04-07; First posted 2022-04-22 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Emergencies; Heart Diseases
Keywords: MEESSI score; ACUTE HEART FAILURE
MeSH Terms: conditions — Emergencies; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MEESSI score — The score aimed to predict the AHF patient's future in the month following management for ED

SUMMARY:
Our primary purpose is to assess MEESSI score in predicting mortality and readmission of patients managed for acute heart failure (AHF) in Emergency Department.

European Society of Cardiology recommend risk stratification for patients with AHF.

DETAILED DESCRIPTION:
Improved risk stratification of acute heart failure (AHF) in the emergency department (ED) may help physicians' decisions regarding patient admission or early discharge disposition. The MEESSI-AHF (Multiple Estimation of risk based on the Emergency department Spanish Score In patients with AHF) score was developed to predict 30-day mortality in patients presenting with AHF EDs in Spain. Whether it performs well in other countries is unknown.

The MEESSI-AHF risk model includes 13 variables readily available on arrival to Emergency Department. The 40% of patients classified as LOW RISK (30-day mortality: <2%) should be considered as potential candidates to be early discharged from Emergency Department without admission after adequate response to initial treatment. The 10% of patients classified as VERY HIGH RISK (30-day mortality: >2%) may clearly benefit from hospital admission.

Objective: To externally validate the MEESSI-AHF score in another country.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient admitted to emergencies with final diagnosis of AHF according to the opinion of two emergency experts after consulting the data from the clinical examination, cardiac echocardiography, and BNP level.
* Subject who accept to participate in the research

Exclusion Criteria:

* Patient who refuse to participate in the study
* Patient with coronary syndrome with ST segment elevation
* Other causes of dyspnea
* Impossibility of giving the patient informed information
* Pregnant woman

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to emergencies with a final diagnosis of AHF
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2009-01-15 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
MEESSI score | 30 days
  predict the AHF patient's future in the month following management in ED with The MEESSI (Multiple Estimation of risk based on the Emergency department Spanish Score In patients with AHF).The MEESSI-AHF risk model includes 13 variables readily available on arrival to Emergency Department. The 40% of patients classified as LOW RISK (30-day mortality: <2%) should be considered as potential candidates to be early discharged from Emergency Department without admission after adequate response to initial treatment. The 10% of patients classified as VERY HIGH RISK (30-day mortality: >2%) may clearly benefit from hospital admission.

SECONDARY OUTCOMES:
Re-admission rate [ Time Frame: 30 days ] | 30 days
  30-day re-admission rate compared between the 4 risk categories defined by the MEESSI score
Mortality rate [ Time Frame: 30 days ] | 30 days
  Mortality rate at 30 days compared between the 4 risk categories defined by the MEESSI score
Sensitivity [ Time Frame: 30 days ] | 30 days
  Sensitivity, specificity and ROC curve of the MEESSI score in relation to the composite criterion according to the 4 risk categories

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Pr, Principal Investigator — University of Monastir
Locations (1):
- Emergency department of University hospital Fattouma Bourguiba, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No
EVALUATE THE PREDICTIVE IMPACT OF THE MEESSI SCORE FOR THE RISK STRATIFICATION OF PATIENTS ADMITTED FOR ACUTE HEART FAILURE IN EMERGENCY STRUCTURES